CLINICAL TRIAL: NCT00646386
Title: Multicenter Study of the Safety and Efficacy of the Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Moderately to Severely Active Psoriatic Arthritis
Brief Title: Study of the Safety and Efficacy of the Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Moderately to Severely Active Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beverly Paperiello/Director, Clinical Development Operations, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-518
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Arthritis; Psoriatic
MeSH Terms: conditions — Arthritis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: adalimumab
- B (Placebo Comparator)
  Interventions: Drug: placebo for adalimumab

INTERVENTIONS:
Drug: adalimumab — 40 mg eow Week 0 - Week 24
  Other Names: ABT-D2E7; Humira
  Arms: A
Drug: placebo for adalimumab — 40 mg eow Week 0 - Week 24
  Other Names: placebo
  Arms: B

SUMMARY:
Multicenter Study of the Safety and Efficacy of the Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects with Moderately to Severely Active Psoriatic Arthritis

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe PsA
* Inadequate response to DMARD therapy
* Corticosteroid stable dose <= 10 mg QD
* DMARDs must have been taken for 3 months and stable dose for 4 weeks
* MTX maximum dose = <= 30 mg/week
* Active chronic plaque PS or documented history of chronic plaque PS

Exclusion Criteria:

* No other active skin disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2003-03; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
ACR20 | Week 12
Adverse Events | Throughout study participation
Sharp Score | Week 24

SECONDARY OUTCOMES:
ACR20, 50, 70 | Weeks 12, 24
Modified Psoriatic Arthritis Response Criteria, HAQ, SF-36, Physician's Global Assessment, PASI, DLQI | Weeks 12 and 24

REFERENCES:
- [Derived] Landewe R, Ritchlin CT, Aletaha D, Zhang Y, Ganz F, Hojnik M, Coates LC. Inhibition of radiographic progression in psoriatic arthritis by adalimumab independent of the control of clinical disease activity. Rheumatology (Oxford). 2019 Jun 1;58(6):1025-1033. doi: 10.1093/rheumatology/key417. PMID 30608620
- [Derived] Mease PJ, Heckaman M, Kary S, Kupper H. Application and modifications of minimal disease activity measures for patients with psoriatic arthritis treated with adalimumab: subanalyses of ADEPT. J Rheumatol. 2013 May;40(5):647-52. doi: 10.3899/jrheum.120970. Epub 2013 Mar 15. PMID 23504383